CLINICAL TRIAL: NCT07081256
Title: A Multicenter, Randomized, Double-blind, Double-dummy, Positive-controlled Phase III Trial, to Evaluate the Efficacy and Safety of QLM2010 for Prevention of Chemotherapy-induced Nausea and Vomiting After Highly Emetogenic Chemotherapy
Brief Title: To Evaluate the Efficacy and Safety of QLM2010 for Prevention of Chemotherapy-induced Nausea and Vomiting After Highly Emetogenic Chemotherapy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QLM2010-301
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-07

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — fosaprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): QLM2010 + dexamethasone
  Interventions: Drug: QLM2010 for injection；dexamethasone
- Treatment group B (Active Comparator): fosaprepitant dimeglumine + palonosetron + dexamethasone
  Interventions: Drug: fosaprepitant dimeglumine for injection；palonosetron hydrochloride injection；dexamethasone

INTERVENTIONS:
Drug: QLM2010 for injection；dexamethasone — QLM2010 for injection；Drug for preventing nausea and vomiting caused by chemotherapy dexamethasone: Drug for preventing nausea and vomiting caused by chemotherapy
  Arms: Treatment group A
Drug: fosaprepitant dimeglumine for injection；palonosetron hydrochloride injection；dexamethasone — fosaprepitant dimeglumine for injection: Drug for preventing nausea and vomiting caused by chemotherapy palonosetron hydrochloride injection: Drug for preventing nausea and vomiting caused by chemotherapy dexamethasone: Drug for preventing nausea and vomiting caused by chemotherapy
  Arms: Treatment group B

SUMMARY:
Compared With Fosaprepitant dimeglumine for Injection and Palonosetron Hydrochloride Injection, to Evaluate the Efficacy and Safety of QLM2010 for Injection for Prevention of Chemotherapy-induced Nausea and Vomiting After Highly Emetogenic Chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide a written informed consent
* 18 years of age or older, of either gender
* Has a diagnosed malignant solid tumor through histological or cytological examination
* Has never been treated with chemotherapy (Antitumor drugs are not used for cancer treatment, or intravesical instillation therapy for bladder cancer is not regarded as chemotherapy)
* Receive the first course of cisplatin-based chemotherapy
* Has a performance status (ECOG scale) of 0 to 2
* Predicted life expectancy of ≥ 3 months

Exclusion Criteria:

* .Subjects with poor blood pressure control after medication
* Subjects with symptomatic brain metastases or any symptoms suggestive of brain metastasis or intracranial hypertension
* Subjects with a history of severe cardiovascular diseases within 3 months prior to the administration of cisplatin, such as acute myocardial infarction, NYHA class II-IV heart failure, etc.
* Subjects with a history of severe torsional ventricular tachycardia, QTcF>480 ms
* Subjects with mental disabilities or severe emotional or mental disorders, The investigators determined that inappropriate for participation in this clinical trial
* Inadequate bone marrow, kidney, and liver function 10. Scheduled to receive any radiation therapy to the abdomen or pelvis from Day -7 through Day 6
* Scheduled to receive moderately or highly emetogenic chemotherapy from Day 2 through Day 6
* Subjects who have experienced emetic events (vomiting or dry vomiting) or nausea within 24 hours before cisplatin-based chemotherapy
* Participated in clinical trials of other drugs within 30 days prior to the administration of cisplatin (received experimental drugs)
* Subjects receiving palonosetron hydrochloride within 21 days before cisplatin-based chemotherapy. Subjects who previously received NK-1 receptor antagonists within 28 days prior to cisplatin-based chemotherapy. Subjects receiving glucocorticoid within 7 days before cisplatin-based chemotherapy.
* Has taken the following agents within the last 48 hours 5-HT3 antagonists, Phenothiazines, Benzamides, Domperidone, Cannabinoids, Benzodiazepines, etc.
* The investigators determined that other conditions were inappropriate for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 665 (Actual)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Complete response during the overall phase after the start of the first cisplatin administration | [Time Frame: 0-120 hours after the start of the first cisplatin administration]
  To compare the rate of subjects achieving and maintaining a complete response (defined as no emetic episode and no need for rescue medication) after the start of the first cisplatin administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhe jiangCancer Hospital, Hangzhou, China